CLINICAL TRIAL: NCT01910506
Title: A Phase 1 Absorption, Metabolism and Excretion Study of [14C]RDEA3170 Orally Administered to Healthy Adult Male Subjects
Brief Title: RDEA3170 AME Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RDEA3170-106
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
MeSH Terms: interventions — verinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RDEA3170 (Experimental)
  Interventions: Drug: RDEA3170 10 mg

INTERVENTIONS:
Drug: RDEA3170 10 mg
  Other Names: RDEA3170 10 mg dose oral solution with 500 μCi of [14C]RDEA3170

SUMMARY:
This study will determine the characteristics of absorption, metabolism, and excretion (AME) of RDEA3170 following a single 10 mg dose of RDEA3170 oral solution with 500 microcuries (µCi) of [14 C]RDEA3170 in healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 50 kg (110 lbs.) and body mass index ≥ 18 and ≤ 30 kg/m2.
* No clinically relevant abnormalities in vital signs, ECG, physical examination or safety laboratory values.
* Screening serum urate level ≤ 7.0 mg/dL.
* Subject has a minimum of 1 bowel movement a day.

Exclusion Criteria:

* History or suspicion of kidney stones.
* History of gastrointestinal ulcers, Helicobacter pylori infection, or other disorders of gastric pH.
* History of previous surgery on the stomach or small intestine (appendectomy is acceptable). Subject has donated blood or experienced significant blood loss (> 450 mL) within 12 weeks prior to Day 1 or has given a plasma donation within 6 weeks prior to Day 1.
* Inadequate venous access or unsuitable veins for repeated venipuncture.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-08; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Characteristics of AME in terms of pharmacokinetics (PK), metabolism, and excretion | Day 1 predose, 15, 30, 45 mins, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 30, 36, 48, 54, 60, 72 hrs postdose (blood and plasma only); Day 1, -12 to 0, 0-6, 6-12, 12-24 hrs postdose (urine and feces only)
  PK profile in terms of AUC, Tmax, Cmax, t1/2, Ae, CLr, and CL/F.
  AUC: area under the concentration-time curve; Tmax: time to reach maximum concentration; Cmax: maximum concentration; t1/2: apparent terminal half-life; Ae: amount of compound excreted in urine unchanged; CLr: renal clearance; CL/F: total body clearance corrected for bioavailability
  Metabolic profile of RDEA3170 in plasma, urine, and feces.
  Excretion in terms of recovery of radioactivity in urine and feces.

SECONDARY OUTCOMES:
Incidence of Adverse Events and Changes in Laboratory, Electrocardiogram, and Vital Signs Parameters | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: S. Baumgartner, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Madison, Wisconsin, United States